CLINICAL TRIAL: NCT04053400
Title: ERASE: Evaluation of the Relationship of the Anesthetic Agent Ketamine and Psychological Sequelae
Brief Title: Evaluating Ketamine and Psychological Sequelae
Acronym: ERASE
Status: Completed | Type: Observational
Sponsor: Defense and Veterans Center for Integrative Pain Management (Other)
Responsible Party: Sponsor
Other Study IDs: 380486
Record Dates: First submitted 2016-01-27; First posted 2019-08-12 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Pain, Ketamine Infusion, Psychologic Sequelae
MeSH Terms: conditions — Pain | interventions — Ketamine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ketamine Group: Active duty military service member injured in theater, AEROVAC-ED out, and received ketamine.
  Interventions: Drug: Ketamine
- Non-Ketamine Comparison Group: Active duty military service member injured in theater, AEROVAC-ED out, and did NOT receive ketamine treatment for pain.

INTERVENTIONS:
Drug: Ketamine
  Groups: Ketamine Group

SUMMARY:
The purpose of this study is to examine the relationship between the use of intravenous infusion of sub-anesthetic dosages of ketamine given for pain to combat casualties and emerging symptoms of Post-Traumatic Stress Disorder (PTSD), depression, anxiety, sleep disruption, and risk of alcohol abuse as identified with behavioral health screening tools. Although ketamine has gained popularity as an analgesic agent, literature related to its psychological impact is sparse.

DETAILED DESCRIPTION:
The purpose of this study is to examine the relationship between the use of intravenous infusion of sub-anesthetic dosages of ketamine given for pain to combat casualties and emerging symptoms of Post-Traumatic Stress Disorder (PTSD), depression, anxiety, sleep disruption, and risk of alcohol abuse as identified with behavioral health screening tools.

This is retrospective case-control study. The data will be analyzed to examine the relationship between exposure to ketamine used as an analgesic agent in combat related trauma care and the expression of psychiatric symptoms measured in the follow-up on the Post Deployment Health Assessment Tool (PDHAT), in use 2003-2007 and the Post Deployment Behavioral Health Assessment (PDBHA), in use 2007 to current date. Coded behavioral health assessment data will be extracted from the research data bank (Protocol IRBnet # 360023, titled "Use of Post Deployment Behavioral Health Assessment Data from Aerovaced Military Admitted to Walter Reed from the Theater of Operations in Iraq and Afghanistan to Establish a Research Data Bank"). This protocol, approved in 2012, has retrospective and prospective components and was designed for studies of this nature. The second objective of this study is to explore demographic and clinical risk factors associated with psychological factors.

Service members who completed the PDHAT or the PDBHA after being AEROVAC-ED from theater for medical care will be grouped according to whether or not they received ketamine for pain before their follow-up assessments. The comparison group for this study will be selected from among those not exposed to ketamine by matching two service members to each in the ketamine group using Injury Severity Scores (ISSs) and Abbreviated Injury Scores (AISs). These scores, originally collected by the US Army Institute of Surgical Research (USAISR) and stored in the Department of Defense Trauma Registry (DoDTR), are an IRB approved addition to the DoP research data bank. WRNMMC and the USAISR have a Memorandum of Understanding allowing use of the scores for research purposes.

ELIGIBILITY:
Inclusion Criteria:

Group I. Ketamine Group

* Active duty military service member injured in theater and treated at WRAMC or at WRNMMC
* 18 years of age or older
* Completed the PBBHA or PDHAT initial and follow up assessment post aerovac from theater
* Received ketamine infusion to treat pain after aero-evacuation for inpatient medical care between Sep 2005 and June 2014
* Received ketamine before completion of the PDHAT or PDBHA follow-up assessment
* ISS scores are available for each individual

Group II. Non-Ketamine Comparison Group

* Active duty military service member injured in theater and treated at WRAMC or at WRNMMC
* 18 years of age or older
* Completed the PBBHA or PDHAT initial and follow up assessment post aerovac from theater
* Did not receive ketamine treatment for pain after aero-evacuation for inpatient medical care before follow-up
* ISS are available for each individual
* Patient will have ISS scores similar to a Ketamine Group patient and a similar timing of injury to the same Ketamine Group patient.

Exclusion Criteria:

* Not treated by WRNMMC/WRAMC hospital staff between Sep 2005 and June 2014
* Not active duty, activated National Guard, or activated Reserve service members
* Younger than 18 years of age
* Did not complete the PDBHA or PDHAT initial and follow-up assessments
* ISS scores are not available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Active military members who were injured in theater and were either treated with ketamine or not.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2014-12; Primary Completion 2017-09 (Actual); Study Completion 2017-09-13 (Actual)

PRIMARY OUTCOMES:
Post Deployment Health Assessment Tool/Post Deployment Behavioral Health Assessment - Coded behavioral health assessment data will be extracted from the research data bank using Injury Severity Scores (ISSs) | 30 days after return home or processing station
  Review wounded warrior's health including mental health post deployment.
Post Deployment Health Assessment Tool/Post Deployment Behavioral Health Assessment - Coded behavioral health assessment data will be extracted from the research data bank using Abbreviated Injury Scores (AISs) | 30 days after return home or processing station
  Review wounded warrior's health including mental health post deployment.

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No